CLINICAL TRIAL: NCT07081295
Title: A Novel Saline-contrast EIT Method for Lung Perfusion Estimation: Without Breath Hold by Low Frequency Band Pass Filter
Brief Title: New Saline-contrast EIT Method Without Breath Hold by Low Pass Filter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: EIT-No breath hold
Record Dates: First submitted 2025-07-02; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No apnea group (Experimental): First, perform the EIT saline contrast method without apnea. After a 10-minute washout period, perform the conventional saline contrast method with apnea.
  Interventions: Other: Injection of hypertonic saline
- Apnea group (Other): First, perform the conventional EIT saline contrast method with apnea. After a 10-minute washout period, perform the saline contrast method without apnea.
  Interventions: Other: Injection of hypertonic saline

INTERVENTIONS:
Other: Injection of hypertonic saline — Injection 10 mL of 10% NaCl through central venous catheter

SUMMARY:
The electrical impedance tomography (EIT) is a bedside, non-invasive, non-radiation imaging tool for lung mornitoring. Currently, the EIT saline-contrast method for lung perfusion evaluation has been widely used in clinical. However, this technique requires the patient to hold breath for 8-30s to avoid the respiratory interference. Hence, it is not suitable for patients that can not tolerate breath hold or unable to maintain a steady apnoea. This study aims to develop an algorithm system based on low frequency band pass filter for EIT saline-contrast lung perfusion estimation without ventilation interruption, and investigate the correlation and agreement of EIT results between the novel method and the conventional breath-hold method.

ELIGIBILITY:
Inclusion Criteria:

* In need of lung perfusion assessment due to clinical condition
* With central venous catheter

Exclusion Criteria:

* Pregnant or breastfeeding females
* contraindications to the use of EIT (automatic implantable cardioverter defibrillator, chest wounds limiting electrode belt placement, implantable pumps, etc.)
* severe hyperchloremia (>155 mmol/L)
* unable to tolerate breath-hold maneuver
* edema disease (nephrotic syndrome, cirrhotic ascites, congestive heart failure, etc.)
* Patients with severe hypernatraemia or hyperchloremia and severe hypertonicity
* Hypertension (>160/100 mmHg), hypokalaemia (> 3.5 mmol/L)
* Acute renal failure in oliguric stage, chronic renal failure with reduced urine output and poor response to diuretics

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Regional V/Q match | Offline analysis, immediately after the saline injection procedure

SECONDARY OUTCOMES:
Pixel-wise lung perfusion fraction | Offline analysis, immediately after the saline injection procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided